CLINICAL TRIAL: NCT02120768
Title: Phase III Study of The Role of Barrier Resection in Local Control in Treatment of Extremity Soft Tissue Sarcomas
Brief Title: Role of Barrier Resection in Local Control for Extremity Recurrent Soft Tissue Sarcomas
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Shi Yingqiang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1310128-1-1312
Record Dates: First submitted 2014-04-01; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Local Recurrence of Malignant Tumor of Soft Tissue
Keywords: Barrier resection; Local recurrence; Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Barrier resection (Experimental): Barrier resection was defined as "en bloc" removal of tumor with surrounding barriers. The barriers include muscular fascia, vascular adventitia, epineurium and periosteum, in some cases where there is no barrier, 3-5cm of healthy tissue is considered equivalent. Barrier resection was developed according to the above characteristics of STSs, which featured with the fact that sarcomas take the path of least resistance and initially grow within the anatomical compartment in which they arose, and the phenomenon that skip metastases are limited within the same anatomic compartment in which the primary lesion is located.Further surgery would be 1cm resection if a recurrence occurs.
  Interventions: Procedure: barrier resection/1cm resection
- 1 cm resection (Active Comparator): Surgical margin width is determined mainly by the distance from the tumor edge to the periphery of the specimen, different margin width of 1-5cm has been recommended for obtaining a safe margin,but the local recurrence rate remains to be 10-25%. Further surgery would be barrier resection if a recurrence occurs.
  Interventions: Procedure: barrier resection/1cm resection

INTERVENTIONS:
Procedure: barrier resection/1cm resection — For Arm "Barrier resection", if a recurrence occurs, patients would be assigned to 1cm resection for their recurrent sarcomas; For Arm "1cm resection", if a recurrence occurs, patients would be assigned to barrier resection for their recurrent sarcomas.

SUMMARY:
The randomized, controlled trial is aiming at comparing local control rate between two surgical resections, barrier resection and local wide resection with 1cm or equivalent normal tissues. This is based on the fact that the goal of local surgical treatment is to remove the tumor with negative margin and best functional outcome, but there is a lack of standard principle of surgery. Some surgical oncologists recommended enlarging surgical field in which case the associated muscle was removed from origin to insertion, the previous surgical scar and radiation field were also grossly remove, though there would be extra trauma and unacceptable function impairment, they believe that patients would benefit from "big operations". Most other surgeons would perform a sarcoma resection through normal tissues, and reported a fair local control as long as a negative margin was obtained. As reported by various authors, recurrent STSs are associated with higher risk to develop further recurrence as compared to primary STSs, thus, efforts should focus on this category of STSs to improve outcome.

DETAILED DESCRIPTION:
1. Background Soft tissue sarcoma (STS) is a category of malignancy with mesenchymal origin, its incidence is 10-20 cases/million and accounts for 1% of all human malignant neoplasms. The most common STSs include undifferentiated polymorphic sarcoma/malignant fibrohistiocytoma (UPS/MFH), synovial sarcoma, fibrosarcoma and liposarcoma.

   The rarity of the tumor, the various subtypes and heterogeneous behavior make the diagnosis and treatment of sarcoma a challenge. Many patients, especially those from developing countries were diagnosed with a late stage disease or recurrent sarcoma being treated with many unplanned resections, which would impact limb function or even survival. Except those with unresectable diseases, surgical resection remains the mainstay of treatment for soft tissue sarcoma, the defined aim of surgery is R0 resection with a good functional outcome. With development of modern strategy and technique, limb sparing surgery has been implied in more than 80% of cases and was proven to have similar local control as amputation without sacrifice of survival. The most common limb sparing surgeries include compartment resection and wide resection. Compartment resection has been gradually replaced by functional compartment resection, aiming at more function preservation, while so far there has been no evidence-based and clinically comprehensible definition of the term "wide resection". Many textbooks still advocate the need to obtain a 2- to 3cm surgical margin width in all directions when resecting a soft tissue sarcoma, but some other orthopaedic and surgical oncologists recommended 1cm or 5cm margin width for STS.

   Local recurrence-free interval is the major end-point in evaluating the quality of surgery, functional outcomes and treatment morbidities are equally important end-points. Five-year local recurrence-free estimations for limb and trunk wall sarcoma should be below 20%, and approaching 10%. Margin status is reported to be a key prognostic factor for local recurrence. Surgical margin width is determined mainly by the distance from the tumor edge to the periphery of the specimen, and should be co-assessed by surgical oncologist and pathologist. Different margin width of 1-5cm has been recommended for obtaining a safe margin, as stated above, but in a limb sparing surgery, margins exceeding 1 cm were obtained in only 47% of patients and it's nearly impossible to obtain 2 cm margins in all directions for an extremity STS. With adjuvant therapies, a close dissection can be adequate in order to preserve important functional structures， but the following questions are unanswered:1. How close is safe for STS resection? 2. Is a margin close to periosteum has the same oncologic result as a margin close to muscular membrane or subcutaneous fat? As we all know that local anatomy influences sarcoma growth by setting natural barriers to extension, and sarcoma might infiltrate or compress surrounding structures, thus, a rational resection should be designed mainly based on the understanding of these characteristics. Scientists investigated different barriers and converted them into different margin width in order to facilitate a safe resection. Among these efforts, a barrier resection was reported to be an option for recurrent extremity STSs and obtained satisfactory local control.

   Barrier resection was defined as "en bloc" removal of tumor with surrounding barriers. The barriers include muscular fascia, vascular adventitia, epineurium and periosteum, in some cases where there is no barrier, 3-5cm of healthy tissue is considered equivalent. Barrier resection was developed according to the above characteristics of STSs, which featured with the fact that sarcomas take the path of least resistance and initially grow within the anatomical compartment in which they arose, and the phenomenon that skip metastases are limited within the same anatomic compartment in which the primary lesion is located. Furthermore, a barrier resection can be designed preoperatively based on imaging studies and is easy to perform intraoperatively based on understanding of local anatomy, and also, it's easy for pathologists to obtain materials for margin evaluation.

   Another content of barrier resection is repair and reconstruction, which includes vessel replacement, dynamic restoration, supporting and wound coverage. With the assistance of repair and reconstruction, sacrifice of margin safety would be no longer needed and in some selected cases, adjuvant radiotherapy would be spared.

   Well defined "R" classification is widely implied to determine the margin status in STSs, in brief, R0 is microscopically negative, R1 is microscopically positive but macroscopically negative, R2 is macroscopically positive. The goal of resection is R0 resection with a good functional outcome, but it's impossible to confirm margin status for all cut edges intraoperatively, while postoperative examination can't guide intraoperative manipulation. So far there has been no evidence-based and clinically comprehensible definition of the term "wide resection", though many guidelines recommended a 1cm normal tissue around tumor. Thus, our study aims at investigating the difference between barrier resection and 1cm margin resection, with local recurrence as main end-point, disease specific survival and functional outcome as secondary end-points.
2. Aims First end-point: Compare the local recurrence between barrier resection and 1cm margin resection.

Secondary end-point:

Disease specific survival (DSS) Functional outcome (MSTS) Surgical complications (Grade)

The first end-point is to compare the local recurrence between barrier resection and 1cm margin resection, it's designed based on the following facts:

1. In compartment theory of Enneking, muscle is independent compartment and most recurrent STSs develop in the same compartment as its original site.
2. The "R" classification of UICC categorized resection margin with margin status, but not margin width, most guidelines recommended 1cm margin resection and a muscle resection from origin to insertion was not required any more. As a result, local control for recurrent STSs was reported to have higher recurrent rate as compared to primary STSs.
3. Some authors in China reported that barrier resection was effective in local control with acceptable extremity functional outcome.

3. Schedule:

From Jan. 2014 to Dec. 2018, as following:

2014.01-2014.03: Methodology and infrastructure construction. 2014.04-2015.09: Sample collection, Surveillance, data gathering. 2015.10-2018.12: Followup, data analysis.

Patients with recurrent extremity STSs are candidates of the study, preoperative CT or MRI should be taken for orientation. As reported previously, barrier resection was associated with comparable local recurrent rate as primary STSs, closing to 15% and 5% of amputation rate, while Eilber reported a recurrent rate and amputation rate for recurrent STSs of 18% and 38%, respectively.

Muscles in trunk don't have independent compartment, thus a barrier resection is not feasible for patients with trunk recurrent STSs. Retroperitoneal STSs have distinctive anatomy and biological behavior, thus are also excluded.

4. Randomization: Patients would be randomized as 1:1 to two groups. Randomization should be taken after radiological evaluation and inclusion. Patients would be stratified according to histologic subtypes and adjuvant therapies.

Patients would be followed up for at least 24 months for disease status and the survival information will be followed up to postoperative 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed recurrent ESTS.
2. Confirmed imaging targets, resectable, no metastasis.
3. No radiochemotherapy in the past 3 months.
4. ECOG status of 0-1.
5. Age between 14 and 80.
6. WBC over 3000/µL，Neutriphil ≥1,500/µL, PLT ≥100,000/µL.
7. Understand the and sign the consent form with compliance.

Exclusion Criteria:

1. Pregnant or lactating.
2. Metastasis.
3. Radiotherapy or chemotherapy in the past 3 months.
4. Another malignancy in the past 3 years.
5. Uncontrollable heart disease or psychologically unstable.
6. Severe infection.
7. In recovery of last operation.
8. Preoperative MSTS score less than 15.
9. Other dysfunctions or situations which assessed to be unsuitable for the trial.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with local recurrence. | up to 2 years

SECONDARY OUTCOMES:
percentage of participants with surgical complications | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chen, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China